CLINICAL TRIAL: NCT02367833
Title: Primary Mechanisms Underlying the Effects of Oral vs. Non-oral Contraceptives on the GH/IGF-1 Axis and Bone Metabolism in Young Women
Brief Title: Effects of Oral vs. Non-oral Contraceptives on the GH/IGF-1 Axis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Massachusetts General Hospital (Other); Purdue University (Other)
Responsible Party: Principal Investigator, Mary Jane DeSouza, Professor of Kinesiology and Physiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000053
Record Dates: First submitted 2015-01-27; First posted 2015-02-20 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Bone; Disorder, Development and Growth
Keywords: Insulin-like growth factor-1; Combined oral contraceptive; Contraceptive Vaginal Ring; Transdermal Contraceptive
MeSH Terms: interventions — Contraceptives, Oral, Combined; Desogestrel; Ortho Evra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Combined Oral Contraceptives (COC) (Experimental): Apri (or generic equivalent - Reclipsen) (30µg/d EE, 150 µg/d desogestrel) is a monophasic dosing regimen of 21 active and 7 placebo pills. On Day 1 of the Intervention, participants in the COC group will begin taking the COC pill. Each participant in this group will ingest active pills from the first pack each day for the first 21 days. Pills ingested on days 22 through 28 are placebo pills. A second pill pack will begin on day 29 and pills with active ingredients will be ingested from the second pack each day for days 29-49. On day 50, the participants will immediately begin a 3rd pill pack, if the post-study testing is still occurring, and will ingest a pill with active ingredients from the third pack for days 50-56 (or for as long as the post-study testing is occurring).
  Interventions: Drug: Combined Oral Contraceptive
- Transdermal Contraceptive (TDC) (Experimental): Participants in the TDC group will apply a 20 cm2 patch (Xulane: 20µg/d EE,150µg/d norelgestromin) to the abdomen, upper arm or buttock. The patch will be changed once weekly on the same day each week for weeks 1-3 (days 1-21, removed on day 22) and weeks 5-8 (days 29-56). Week 4 (days 22-28) will be a patch-free week. As soon as the post-study testing is complete, subjects will remove the patch.
  Interventions: Drug: Transdermal Contraceptive
- Contraceptive Vaginal Ring (CVR) (Experimental): Participants in the CVR group (NuvaRing - 15µg/d EE/120µg/d etonogestrel) will insert a vaginal ring into the vagina on Day 1 of the intervention. The vaginal ring will be removed and discarded after 3 weeks of continuous use (days 1-21 of continuous use and removed on day 22). There will be one week (days 22-28) that will be ring-free. A new ring will be inserted for days 29-49. On day 50, the second ring will be removed, and a third ring will be immediately inserted into the vagina (if the post-study testing is still occurring). The third ring will remain in the vagina for the last week of the post-study period (days 50-56). As soon as the post-study testing is complete, subjects will remove the ring.
  Interventions: Drug: Contraceptive Vaginal Ring
- Control Group (No Intervention): The Control group will complete all procedures with the exception of contraceptive therapy.

INTERVENTIONS:
Drug: Combined Oral Contraceptive — The proposed study is a preclinical, multi-site trial comparing the short-term effects of oral and non-oral ethinyl estradiol on the GH/IGF-1 axis and bone metabolism. Using a prospective repeated measures design, we will test the effects of 2 cycles of combined oral contraceptive (Apri or Reclipsen) on the GH/IGF-1 axis.
  Other Names: Apri (Reclipsen)
  Arms: Combined Oral Contraceptives (COC)
Drug: Transdermal Contraceptive — The proposed study is a preclinical, multi-site trial comparing the short-term effects of oral and non-oral ethinyl estradiol on the GH/IGF-1 axis and bone metabolism. Using a prospective repeated measures design, we will test the effects of 2 cycles of a transdermal contraceptive (Xulane) on the GH/IGF-1 axis.
  Other Names: Xulane
  Arms: Transdermal Contraceptive (TDC)
Drug: Contraceptive Vaginal Ring — The proposed study is a preclinical, multi-site trial comparing the short-term effects of oral and non-oral ethinyl estradiol on the GH/IGF-1 axis and bone metabolism. Using a prospective repeated measures design, we will test the effects of 2 cycles of vaginal ring contraceptive (Nuva Ring) on the GH/IGF-1 axis.
  Other Names: Nuva Ring
  Arms: Contraceptive Vaginal Ring (CVR)

SUMMARY:
This study will determine whether the negative effects of combined oral contraceptive (COC) therapy on the growth hormone/insulin-like growth factor-1 (GH/IGF-1) axis and bone turnover are dependent on the route of administration such that an attenuation of these effects is observed when a comparable dose of non-oral transdermal contraceptive (TDC) and contraceptive vaginal ring therapy (CVR) are also tested.

DETAILED DESCRIPTION:
This study is a preclinical, multi-site trial (Penn State University and Purdue University) that will determine whether the negative effects of combined oral contraceptive (COC) therapy on bone turnover are dependent on the route of administration such that an attenuation of these effects is observed when a comparable dose of non-oral transdermal contraceptive (TDC) therapy and contraceptive vaginal ring (CVR) therapy are also tested. Millions of women use COC therapy for birth control purposes or regulation of menstrual cycles. TDC and CVR therapies are relatively new FDA-approved contraceptive alternatives to COC. The purpose of the proposed project is to address the potential mechanism(s) by which oral ethinyl estradiol (EE) may negatively impair bone via "first pass" effects on the liver and compare these effects to transdermally-administered and vaginally-administered EE in young women. We will assess mechanistic effects by way of 2-day serial sampling and by an insulin-like growth factor (IGF-1) generation test. The IGF-1 generation test was developed over 20 years ago and is currently used to diagnose growth hormone (GH) insensitivity. IGF-1 generation tests may also be used to amplify effects not observable by the assessment of fasting or serial concentrations of systemic IGF-1(secreted by the liver) and its associated binding proteins. This study will be the first study to examine the physiological mechanisms whereby the route of estrogen administration affects the GH/IGF-1 axis and bone turnover in young women.

The overall purpose of this study is to explore differences in liver metabolism and bone turnover of oral versus transdermal and vaginal contraceptive therapy. In an effort to expose the route-dependent effects of oral versus transdermal and vaginal contraceptive therapy on liver and bone metabolism, we will examine the effects of ethinyl estradiol on serially-assessed fasting concentrations of the GH/IGF-1 axis and bone turnover and explore physiological mechanisms underlying hepatic responsiveness to oral versus transdermal and vaginal contraceptive therapy using an IGF-1 Generation Test as a probe.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18-30 yrs
3. BMI 18-29 kg/m2
4. Non-smoking
5. Not using hormonal contraceptives for at least 6 months prior
6. Not currently pregnant nor intending to become pregnant in the next 6 months
7. Not lactating
8. No apparent metabolic, endocrine, musculoskeletal, or severe psychiatric disease
9. Willing to adhere to maintenance of current exercise training and diet and remain weight stable (±2 kg) during study
10. Variable physical activity acceptable, but mode must be primarily weight bearing
11. At least 9 menses in past 12 months
12. Willing to quit taking any current nutritional supplements and take Calcium and Vitamin D supplements for the duration of the study.
13. If 21 or older, a normal Pap smear must be confirmed.

Exclusion Criteria:

1. Non-weight bearing exercise as primary mode of physical activity
2. Known or suspected metabolic or endocrine disease
3. Pregnant
4. Currently consuming large amounts of soy products
5. Regular consumption of grapefruit juice
6. Current clinical eating disorder or other axis 1 psychiatric or bipolar disorders
7. Oral or hormonal contraceptive use in the last 6 months
8. Currently amenorrheic
9. Hyperparathyroidism
10. Liver or renal disease
11. Evidence of malabsorption or skeletal disorder
12. Thyroid abnormalities (controlled hypothyroidism acceptable)
13. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDS)
14. Taking medications known to have interactions with contraceptive therapy
15. Division I Athlete, on or off season
16. Other Exclusion Criteria proposed by the World Health Organization COC Contraindications (Grossman, 2011)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane De Souza, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- Women's Health and Exercise Laboratories, The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Grossman D, White K, Hopkins K, Amastae J, Shedlin M, Potter JE. Contraindications to combined oral contraceptives among over-the-counter compared with prescription users. Obstet Gynecol. 2011 Mar;117(3):558-565. doi: 10.1097/AOG.0b013e31820b0244. PMID 21343758
- [Derived] Allaway HCM, Misra M, Southmayd EA, Stone MS, Weaver CM, Petkus DL, De Souza MJ. Are the Effects of Oral and Vaginal Contraceptives on Bone Formation in Young Women Mediated via the Growth Hormone-IGF-I Axis? Front Endocrinol (Lausanne). 2020 Jun 16;11:334. doi: 10.3389/fendo.2020.00334. eCollection 2020. PMID 32612574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Penn State University and Purdue University campuses from January 2015 to June 2016.
Pre-assignment Details: A total of 60 participants enrolled in the study and 34 participants did not pass the screening phase.
Period: Overall Study
Arm/Group | Combined Oral Contraceptives (COC) | Contraceptive Vaginal Ring (CVR) | Control Group
Started | 9 | 9 | 8
Completed | 8 | 8 | 8
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Combined Oral Contraceptives (COC) | Contraceptive Vaginal Ring (CVR) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Full Range); unit: years] | 23.6 [20 to 28] | 22.3 [18 to 29] | 23.1 [19 to 30] | 23 [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 24
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 5 | 5 | 5 | 15
  Asian | 1 | 1 | 0 | 2
  African American/Black | 0 | 0 | 1 | 1
  Latin American | 0 | 0 | 1 | 1
  Other | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Changes in Insulin-like Growth Factor-1 (IGF-1), IGF Binding Proteins (IGFBP-1, IGFBP-3), and Acid Labile Subunit (ALS)
Description: Changes in serially-sampled fasting serum concentrations of insulin-like growth factor-1 (IGF-1) before and after 49 days of contraceptive therapy. Data were only collected for IGF-1 levels, no assays were performed for IGFBP-1, IGFBP-3, and acid labile subunit (ALS) and no raw data were collected due to insufficient funds.
Time Frame: Baseline and post-49 days of contraceptive therapy
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Control Group | Combined Oral Contraceptives (COC) | Contraceptive Vaginal Ring (CVR)
Number analyzed (Participants) | 8 | 8 | 8
ng/mL
  Baseline IGF-1 Concetration | 220.6 (14.8) | 228.7 (13.6) | 197.1 (15.2)
  Post-Therapy IGF-1 Concentration | 221.4 (11.5) | 185.9 (10.3) | 175.2 (11.1)

2. Secondary Outcome: Changes in Bone Turnover Markers
Description: Changes in serially-sampled fasting serum concentrations of markers of bone formation (osteocalcin, P1NP) and bone resorption (NTx, and CTx) before and after contraceptive therapy.
Time Frame: Baseline and post-49 days of contraceptive therapy
Population: No data was collected due to insufficient funds.
Arm/Group | Control Group | Combined Oral Contraceptives (COC) | Contraceptive Vaginal Ring (CVR)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Changes in GH-stimulated IGF-1 Secretion
Description: Changes in IGF-1, IGFBP-1, IGFBP-3,and ALS in response to exogenously administered GH before and after contraceptive therapy.
Time Frame: 49 days of contraceptive therapy
Population: No data was collected due to insufficient funds.
Arm/Group | Control Group | Combined Oral Contraceptives (COC) | Contraceptive Vaginal Ring (CVR)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during period of study enrollment through study completion, a period of approximately 4 months.
Arm/Group | Control Group | Combined Oral Contraceptives (COC) | Contraceptive Vaginal Ring (CVR)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02367833/Prot_SAP_000.pdf